CLINICAL TRIAL: NCT02606344
Title: Effect of a Micro-finance-based Intervention for the Prevention of Intimate-partner Violence and HIV: a Multi-centric Randomized Trial
Brief Title: Effect of a Micro-finance-based Intervention for the Prevention of Intimate-partner Violence and HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Sonal Foundation, India (Other); Vinita Nursing Home, India (Other); Macmillan Research Group UK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: nmp/22186
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: HIV; AIDS; Domestic Violence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (IG) (Experimental): Loans were provided to poor women who enrolled in the intervention group. A participatory learning and action curriculum was integrated into loan meetings, which took place every 2 weeks.
  Interventions: Other: Mico-finance based intervention
- Control Group (CG) (No Intervention)

INTERVENTIONS:
Other: Mico-finance based intervention
  Arms: Intervention Group (IG)

SUMMARY:
The high rates of HIV infection in women have brought into sharp focus the problem of violence against women. There is a growing recognition that women and girls' risk of and vulnerability to HIV infection is shaped by deep-rooted and pervasive gender inequalities violence against them in particular. The links between intimate partner violence and HIV/AIDS are explained by biological as well as sociocultural and economic factors.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old;
* Must plan to reside in study areas for the next 12 months
* Must visit camp at least 1 time per week
* Must provide contact information of friend or family member

Exclusion Criteria:

* Unwilling to provide local information
* Psychological disturbance, cognitive impairment or threatening behavior

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of New Sexually Transmitted Infections | 12 months

SECONDARY OUTCOMES:
Proportion of women Reporting Physical, Sexual, or Psychological Partner Violence | 12 Months
Proportion of unprotected sexual acts with partner | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Kalvinder Kour, MBA, Principal Investigator — NMP Medical Research Institute, India; Neha Sharma, PhD, Study Director — Macmillan Research Group UK; Vinita Makkad, MD, Principal Investigator — Vinita Nursing Home, India
Locations (3):
- India (3):
  - Sonal Foundation, Mahesāna, Gujarat
  - Vinita Nursing Home, Hindaun, Rajasthan
  - NMP Medical Research Institute, Deharadun, Uttarakhand